CLINICAL TRIAL: NCT04489017
Title: Palmitoylethanolamide Combined With Luteoline in Frontotemporal Dementia Patients. A Randomized Controlled Trial
Acronym: PEA-FTD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SPE.107
Record Dates: First submitted 2020-04-13; First posted 2020-07-28 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2022-06

CONDITIONS: Frontotemporal Dementia
Keywords: dopamine; frontal cortex; GABA
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEA-LUT (Experimental): PEA-LUT administration at the oral dosage of 700 mg x 2/day for 24 weeks
  Interventions: Dietary Supplement: PEA-LUT
- PLACEBO (Placebo Comparator): PLACEBO administration at the oral dosage of 700 mg x 2/day for 24 weeks
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: PEA-LUT — PEA-LUT administration at the oral dosage of 700 mg x 2/day
  Arms: PEA-LUT
Dietary Supplement: PLACEBO — PLACEBO administration at the oral dosage of 700 mg x 2/day
  Arms: PLACEBO

SUMMARY:
Frontotemporal dementia (FTD) is a devastating neurodegenerative disorder. It is the second most frequent cause of presenile neurodegenerative dementia in those less than 65 years of age. Currently, there is no effective pharmacological treatment to slow down the progression of FTD. Recently, it has been proposed that neuroinflammation could be involved in specific forms of FTD and that novel drugs targeting neuroinflammation could potentially be useful in FTD treatment. An available form of ultra-micronized PEA combined with luteoline (PEA-LUT) has gained attention for its proven anti-inflammatory and neuroprotective properties reported in neurodegenerative conditions related to FTD, such as Amyotrophic Lateral Sclerosis. The administration of PEA-LUT treatment may have a clinical impact in behavioural variant FTD (bv-FTD) patients. In particular, PEA-LUT treatment could be able to reduce behavioural disturbances, the more disabling symptoms in bv-FTD, with a related improvement of daily living activities of affected people. Moreover, a multimodal approach (cognitive/neurophysiological) can be used to assess the brain correlates related to the clinical improvement associated with PEA-LUT treatment, thus making remarkable strides in understanding how FTD affects the brain. Potentially the proposed project could provide a valid treatment for cognitive and behavioural dysfunction in FTD patients, with consistent impact for the National Health Systems and minimum cost for the patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of probable Frontotemporal dementia behavioural variant (bv-FTD) based on the International consensus clinical diagnostic criteria described by Rascovsky et al., 2011.
2. The patient is a man or a woman, aged from 40 to 85 years.
3. The patient has a Clinical Dementia Rating-FTD (CDR-FTD) total score of ≤2 at Screening.
4. The patient has not been treated with acetylcholinesterase inhibitor (AChEI), i.e., donepezil, galantamine, or rivastigmine, at the time of screening.
5. The patient is able to comply with the study procedures in the view of the investigator.
6. Evidence of frontotemporal hypometabolism at PET imaging.
7. Evidence of amyloid markers excluding Alzheimer's disease (cerebrospinal fluid Abeta/Tau dosages or amyloid PET imaging).

Exclusion Criteria:

1. Significant neurodegenerative disorder of the central nervous system other than FTD e.g., Alzheimer's disease, Lewy body dementia, Parkinson's disease, multiple sclerosis, progressive supranuclear palsy, normal pressure hydrocephalus, Huntington's disease, any condition directly or indirectly caused by Transmissible Spongiform Encephalopathy (TSE), Creutzfeldt-Jakob Disease (CJD), variant Creutzfeldt-Jakob Disease (vCJD), or new variant Creutzfeldt-Jakob Disease (nvCJD)
2. Significant intracranial focal or vascular pathology seen on brain MRI scan within a maximum of 6 months before Baseline leading to a diagnosis other than probable FTD.
3. The patients has history of seizure (with the exception of febrile seizures in childhood).
4. Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MR imaging.
5. Treatment currently or within 3 months before Baseline with any of the following medications: Typical and Atypical antipsychotics (i.e., Clozapine, Olanzapine); Antiepileptics drugs (i.e., Carbamazepine, Primidone, Pregabalin, Gabapentin); Antidepressants (i.e., Citalopram, Duolxetine, Paroxetine).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating Scale- Frontotemporal dementia Sumo of Boxes (CDR-FTD-SOB) | 24 weeks
  Battery to evaluate global disease severity

SECONDARY OUTCOMES:
Frontal Assessment Battery (FAB) | 24 weeks
  Battery to evaluate executive functions
Screening for aphasia in Neurodegeneration (SAND) | 24 weeks
  battery to evaluate language functions
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 24 weeks
  battery to evaluate activities of daily living
Mini Mental State Examination (MMSE) | 24 weeks
  battery to evaluate global cognition
Long intracortical inhibition (LICI) | 24 weeks
  TMS protocol to evaluate GABA(B)ergic transmission
Sort intracortical inhibition (SICI) | 24 weeks
  TMS protocol to evaluate GABA(B)ergic transmission
TMS-EEG | 24 weeks
  power in beta-gamma band to evaluate prefrontal cortical oscillatory activity
Neuropsychiatric Inventory (NPI) | 24 weeks
  Battery to assess behavioral changes
Addenbrooke's Cognitive Examination Revised (ACE-R) | 24 weeks
  Battery to evaluate global cognition changes
Frontal Behavioural Inventory | 24 weeks
  Battery to evaluate behavioural functions

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Giacomo Koch, Rome
  - Santa Lucia Foundation, Rome

IPD SHARING:
Plan to Share IPD: Undecided